CLINICAL TRIAL: NCT06554938
Title: Efficacy of Dental Hygiene Aids in Reducing Gingival Bleeding and Plaque Among Orthodontic Patients. A Randomized Controlled Trial
Brief Title: Efficacy of Dental Hygiene Aids in Reducing Gingival Bleeding and Plaque Among Orthodontic Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajman University (Other)
Responsible Party: Principal Investigator, sudhir rama varma, Clinical Assistant Professor, Ajman University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: D-F-H-31-Oct-ii
Record Dates: First submitted 2024-08-09; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Gingival Bleeding; Dental Plaque
Keywords: Dental plaque; Gingival Bleeding; Oral irrigator; waterpik; super floss
MeSH Terms: conditions — Gingival Hemorrhage; Dental Plaque | interventions — Dental Devices, Home Care

STUDY DESIGN:
Intervention Model Description: The study comprised 18-35-year-old girls and boys planning orthodontic treatment. Participants had upper right tooth to lower left molar braces, a pocket depth of 3 mm, and had not flossed in 24 hours. Smoking, periodontal disease, missing teeth, voids between teeth in the arch, and systemic disorders disqualified participants.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomized trial by lots
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- water pik (Active Comparator): One side of the mouth was flossed with Super Floss® (Oral-B) and the other with Waterpik®.
  Interventions: Device: water pik
- Super floss (Active Comparator): One side of the mouth was flossed with Super Floss® (Oral-B) and the other with Waterpik®.
  Interventions: Device: Super floss

INTERVENTIONS:
Device: water pik — One side of the mouth was flossed with Super Floss® (Oral-B) and the other with Waterpik®.
  Other Names: oral irrigator
  Arms: water pik
Device: Super floss — One side of the mouth was flossed with Super Floss® (Oral-B) and the other with Waterpik®.
  Other Names: Dental floss
  Arms: Super floss

SUMMARY:
Adult orthodontic patients aged 18-30 were included in a randomised, single-blind clinical research using a split-mouth design at a dental clinic. Both the Waterpik® and the Super-Floss® water flossers are manufactured by Oral-B.

DETAILED DESCRIPTION:
In order to reduce gingival inflammation and remove subgingival plaque, oral hygiene therapy is necessary. The available evidence indicates that mechanical plaque control, which patients administer themselves daily, is the most important factor in managing and reducing plaque accumulation.

Aim: This research aimed to determine whether Waterpik or Superfloss was more effective in lowering the gingival bleeding score and plaque.

Methods: Adult orthodontic patients aged 18-30 were included in a randomised, single-blind clinical research using a split-mouth design at a dental clinic. Both the Waterpik® and the Super-Floss® water flossers are manufactured by Oral-B.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18-35 years undergoing orthodontic treatment and
* systemically healthy without habits

Exclusion Criteria:

* Participants not undergoing orthodontic treatment and participants undergoing orthodontic treatment in the included age category but with systemic conditions prevalent
* missing teeth and
* treated previously for periodontal conditions

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Gingival bleeding | 24 to 72 hours; 24 hours means at baseline and 72 hours is post intervention
  Gingival bleeding scores will be evaluted
Dental plaque | 24 to 72 hours; 24 hours means at baseline and 72 hours is post intervention
  Dental plaque scores will be evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Ajman University, Ajman, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
study protocol, Data and statistical analysis
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be shared when requested
Access Criteria: The data can be shared by Email